CLINICAL TRIAL: NCT02668107
Title: Electromyographic Activity of Preterm Newborns Submitted to Hammock Positioning : a Randomized Clinical Trial
Brief Title: Electromyographic Activity of Preterm Newborns Submitted to Hammock Positioning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Principal Investigator, Isabel Cristina de Almeida Eyre, Mrs, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CAAE 43874915.0.0000.5201
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Infant, Premature, Diseases
MeSH Terms: conditions — Infant, Premature, Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Hammock positioning) (Active Comparator): Babies in the intervention group (IG), will be positioned supine in a hammock in the incubator, with the appropriate postural adjustments.
  Interventions: Other: Hammock positioning
- Control Group (No Intervention): Those selected for the control group (CG) will be placed in the incubator following the service routine.

INTERVENTIONS:
Other: Hammock positioning — Babies in the intervention group (IG), will be positioned supine in a hammock(hammock positioning) in the incubator, with the appropriate postural adjustments.
  Arms: Intervention Group (Hammock positioning)

SUMMARY:
To compare and analyze the effects on the electromyographic activity of preterm newborns placed in the hammock position with the activity of newborns not placed in this position.

DETAILED DESCRIPTION:
Randomized clinical trial, according to CONSORT standards, with newborn preterm gestational age <34 weeks and birth weight <1500 g, admitted to the intensive care unit. Newborns will be randomized. Those selected for the control group (CG) will be placed in the incubator following the service routine. Babies in the intervention group (IG), will be positioned supine in a hammock in the incubator, with the appropriate postural adjustments. The evaluation of muscle activity will be carried out through surface electromyography. Evaluations shall be performed immediately before the intervention; immediately after 24 hours of intervention; and within 24 hours without intervention, in order to compare the values before and after the intervention of the two groups, as well as if the effects of the intervention are maintained after its removal.

ELIGIBILITY:
Inclusion Criteria:

* Preterm Infants with gestational age <34 weeks
* Free from mechanical ventilation in the last 48 hours prior to electromyographic evaluation
* Not in use of supplemental oxygen at the time of assessment

Exclusion Criteria:

* Apgar score of less than seven in the fifth minute
* Previous history of perintraventricular hemorrhage grade III and / or IV
* Congenital infection
* Congenital heart defects
* Neonatal Obstetric traumas
* Gastroesophageal Reflux Disease
* Genetic syndromes
* Congenital malformations
* Sepsis with meningitis
* Orthopedic and musculoskeletal alterations

Ages: 1 Day to 20 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2015-08; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Increase in Muscle activity | 24 hours
  In preterm infants placed in hammocks with gestational age less than or equal to 34 weeks and birth weight less than or equal to 1500g:
  1. Muscle activity of the elbow flexors (corresponding to the biceps muscle) and knee flexors (corresponding mainly to the hamstring muscle group) increases.
  2. The increase in electromyographic activity persists 24 hours after removal of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Eyre, Bachelor, Principal Investigator — Instituto de Medicina Integral Professor Fernando Figueira
Locations (1):
- Instituto de Medicina Integral Professor Fernando Figueira, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No